CLINICAL TRIAL: NCT01202669
Title: Heart Rate Changes in Subjects With Epilepsy During an Epilepsy Monitoring Unit Admission
Brief Title: Heart Rate Changes in Subjects With Epilepsy
Status: Completed | Type: Observational
Sponsor: Cyberonics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: E-30
Record Dates: First submitted 2010-08-06; First posted 2010-09-16 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Epilepsy patients, EMU stay
  Interventions: Other: No intervention planned, observational study only.

INTERVENTIONS:
Other: No intervention planned, observational study only. — No intervention planned, observational study only.

SUMMARY:
The purpose of this study is to collect continuous observational data during a clinical Epilepsy Monitoring Unit evaluation.

DETAILED DESCRIPTION:
Observational, unblinded, non-randomized, multisite study designed to collect data on up to 500 subjects undergoing evaluation for epilepsy in EMUs. Subjects currently enrolled or that previously participated in this study may be eligible for the E-30-S sub-study.

ELIGIBILITY:
Inclusion Criteria:

Patients enrolled in the study must meet all of the following criteria:

1. Patient has a clinical diagnosis of epilepsy requiring evaluation in an epilepsy monitoring unit (EMU).
2. Patient likely requires an EMU evaluation for a period of at least 24 hours.
3. Patient is currently taking at least one antiepileptic medication.
4. Patient must be in good general health and fully ambulatory.
5. Patient or guardian must be willing and able to complete informed consent/assent and HIPAA authorization.

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible to be enrolled in the study:

1. Patients with severe psychiatric disease that in the investigator's judgment would prevent the patient's successful completion of the study.
2. Patients with a history of status epilepticus.
3. Patients prescribed drugs specifically for a cardiac or autonomic disorder that in the investigator's opinion would affect heart rate response. Drugs with secondary cardiac or autonomic actions are allowed.
4. Patients with cardiovascular arrhythmias or cardiac disease that would preclude the ability to detect intrinsic changes in heart rate due to exercise, stress, or seizure. This would include but not be limited to chronic atrial fibrillation, chronotropic incompetence, and permanent cardiac pacemaker implantation.
5. Patients with a history of dependence on alcohol or narcotic drugs within the past 2 years as defined by DSM IV-R.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Epilepsy patients indicated for epilepsy monitoring unit stay.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2010-08; Primary Completion 2012-10 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Collection of physiologic data during an Epilepsy Monitoring Unit (EMU) stay | up to 7 days
  To collect continuous observational video, electroencephalogram (EEG), electrooculogram (EOG), and electrocardiogram (ECG) data during ictal and non-ictal events occurring over a clinical EMU evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Olin, Study Director — Employee
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - University of Chicago, Chicago, Illinois

REFERENCES:
- [Background] VAN BUREN JM. Some autonomic concomitants of ictal automatism; a study of temporal lobe attacks. Brain. 1958 Dec;81(4):505-28. doi: 10.1093/brain/81.4.505. No abstract available. PMID 13618449
- [Background] Marshall DW, Westmoreland BF, Sharbrough FW. Ictal tachycardia during temporal lobe seizures. Mayo Clin Proc. 1983 Jul;58(7):443-6. PMID 6865478
- [Background] Keilson MJ, Hauser WA, Magrill JP. Electrocardiographic changes during electrographic seizures. Arch Neurol. 1989 Nov;46(11):1169-70. doi: 10.1001/archneur.1989.00520470023018. PMID 2818251
- [Background] Smith PE, Howell SJ, Owen L, Blumhardt LD. Profiles of instant heart rate during partial seizures. Electroencephalogr Clin Neurophysiol. 1989 Mar;72(3):207-17. doi: 10.1016/0013-4694(89)90245-9. PMID 2465123
- [Background] Schernthaner C, Lindinger G, Potzelberger K, Zeiler K, Baumgartner C. Autonomic epilepsy--the influence of epileptic discharges on heart rate and rhythm. Wien Klin Wochenschr. 1999 May 21;111(10):392-401. PMID 10413832
- [Background] Di Gennaro G, Quarato PP, Sebastiano F, Esposito V, Onorati P, Grammaldo LG, Meldolesi GN, Mascia A, Falco C, Scoppetta C, Eusebi F, Manfredi M, Cantore G. Ictal heart rate increase precedes EEG discharge in drug-resistant mesial temporal lobe seizures. Clin Neurophysiol. 2004 May;115(5):1169-77. doi: 10.1016/j.clinph.2003.12.016. PMID 15066542
- [Background] Leutmezer F, Schernthaner C, Lurger S, Potzelberger K, Baumgartner C. Electrocardiographic changes at the onset of epileptic seizures. Epilepsia. 2003 Mar;44(3):348-54. doi: 10.1046/j.1528-1157.2003.34702.x. PMID 12614390
- [Background] Novak V, Reeves AL, Novak P, Low PA, Sharbrough FW. Time-frequency mapping of R-R interval during complex partial seizures of temporal lobe origin. J Auton Nerv Syst. 1999 Sep 24;77(2-3):195-202. PMID 10580303
- [Background] Epstein MA, Sperling MR, O'Connor MJ. Cardiac rhythm during temporal lobe seizures. Neurology. 1992 Jan;42(1):50-3. doi: 10.1212/wnl.42.1.50. PMID 1734323
- [Background] Zijlmans M, Flanagan D, Gotman J. Heart rate changes and ECG abnormalities during epileptic seizures: prevalence and definition of an objective clinical sign. Epilepsia. 2002 Aug;43(8):847-54. doi: 10.1046/j.1528-1157.2002.37801.x. PMID 12181003
- [Background] van Elmpt WJ, Nijsen TM, Griep PA, Arends JB. A model of heart rate changes to detect seizures in severe epilepsy. Seizure. 2006 Sep;15(6):366-75. doi: 10.1016/j.seizure.2006.03.005. Epub 2006 Jul 7. PMID 16828317